CLINICAL TRIAL: NCT01824797
Title: Determining Changes in Bone Metabolism After Bariatric Surgery in Postmenopausal Women
Brief Title: Bone Metabolism After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00044248
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Osteoporosis
Keywords: Bone mineral density; sleeve gastrectomy; roux-en-y; postmenopausal females; bone loss
MeSH Terms: conditions — Obesity; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be collected from the subjects preoperatively and 12 months postoperatively. The serum will be used at the completion of the study to run enzyme-linked immunosorbent assay (ELISA) to determine biochemical changes in their bone metabolism.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Roux-en-Y Gastric Bypass: Changes in bone mineral density will be determined by comparing a peroperative DEXA scan with a one year postoperative DEXA scan on postmenopausal subjects who have already planned to undergo Roux-en-Y gastric bypass or sleeve gastrectomy. Serum will be collected from subjects preoperatively and 12 months postoperatively. The serum will be used at the completion of the study to run enzyme-linked immunosorbent assay (ELISA) to determine biochemical changes in bone metabolism.
- Sleeve Gastrectomy: Changes in bone mineral density will be determined by comparing a peroperative DEXA scan with a one year postoperative DEXA scan on postmenopausal subjects who have already planned to undergo Roux-en-Y gastric bypass or sleeve gastrectomy. Serum will be collected from subjects preoperatively and 12 months postoperatively. The serum will be used at the completion of the study to run enzyme-linked immunosorbent assay (ELISA) to determine biochemical changes in bone metabolism.

SUMMARY:
The purpose and objective of this study is to determine the changes in bone metabolism after bariatric surgery in postmenopausal women.

This is a prospective cohort study that will enroll up to 40 postmenopausal female subjects with class II and III obesity from the Duke Center for Metabolic and Weight Loss Surgery. The study team will enroll subjects that are already being scheduled for either sleeve gastrectomy or Roux-en-Y gastric bypass. The osteoclast activity, the osteoblast activity, and the bone mineral density will be measured in all subjects preoperatively and 12 months postoperatively through research specific blood tests and Dual energy x-ray Absorptiometry (DEXA) scans.

The primary endpoints are change in osteoclast activity as measured by C-terminal telopeptide of type I collagen and change in bone density as measured by DEXA scan. These are continuous variable and given the small sample size the investigators will use a nonparametric Wilcoxon rank-sum test to compare the difference in one year change in these variables. There is a slight risk of loss of confidentiality. Every effort will be made to protect all PHI. There is also the risk of increased exposure to radiation from the DEXA scans performed twice with each subjects participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women as determined by having a history of no menstrual bleed for greater than one year.
2. Body Mass Index ≥35 kg/m² and stable weight for the previous 3 months.
3. Able to speak and read English.
4. Being scheduled for either Roux-en-Y gastric bypass or sleeve gastrectomy.

Exclusion Criteria:

1. A documented history of osteoporosis or currently receiving medical treatment for osteoporosis with bisphosphonates, teriparatide, raloxifene, or denosumab.
2. Weight greater than 295 pounds as this is the weight limit for our Dual-energy X-ray absorptiometry machine.
3. Current or past (less than 1 year from enrollment) usage of estrogen hormone replacement therapy.
4. Current smoker
5. Any history of glucocorticoid use greater than one year in duration or current use of glucocorticoids.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal females scheduled to undergo Roux-en-Y gastric bypass or Sleeve Gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Bone Mineral Density | Baseline to one year postoperative
  Changes in bone mineral density will be determined by comparing a peroperative DEXA scan with a one year postoperative DEXA scan on postmenopausal subjects who have already planned to undergo Roux-en-Y gastric bypass or sleeve gastrectomy.

SECONDARY OUTCOMES:
Biochemical Changes in Bone Metabolism | Baseline to one year postoperative
  Serum will be collected from the subjects preoperatively and 12 months postoperatively. The serum will be used at the completion of the study to run enzyme-linked immunosorbent assay (ELISA) to determine biochemical changes in their bone metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Guerron, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Metabolic and Weight Loss Surgery, Durham, North Carolina, United States

REFERENCES:
- See also: Luhrs, A.R., Davalos, G., Lerebours, R. et al. Surg Endosc (2019) — https://doi.org/10.1007/s00464-019-06922-8